CLINICAL TRIAL: NCT06710886
Title: The Effect of Listening to Calming Music
Brief Title: Listening to Calming Music
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB202401783
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: Music; Autonomic State
Keywords: Polyvagal Theory; Adversity; Relaxation

STUDY DESIGN:
Intervention Model Description: In Phase 1: The participants will listen to the brief music demo together after completing the pre-assessment. After the demo is completed, participants will listen to the 15-minutes of music. For those who opt out of listening to the 15-minutes of music, they will be asked to complete the post-assessment. Following the 15-minute music session, the remaining participants will be asked to complete the post-assessment.
  In Phase 2: Participants will be randomly assigned to the augmented or control music group. Both groups will complete a pre-survey and provide a saliva sample. Then, they will be equipped with a HR band (polar exercise band) and baseline HR will be established within 5 minutes. Following the 15-minutes of music, participants will provide 5 minutes of HR information post-intervention, provide a saliva sample, and complete a post-survey.
Who Masked: Participant
Masking Description: Phase 2: Participants will be randomly assigned via a random number generator to either the augmented group or the control group. The participant will be blinded to the group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Theme (Experimental): In phase 1:
  Participants complete the pre-survey. After that, the participants will listen to a brief demo followed by the 15-minutes of augmented music. After completion of the music, the participants will complete the post-survey.
  In phase 2:
  Participants complete the pre-survey, and provide 1.5-2mL of saliva. Then, they will be equipped with a HR band (polar exercise band). After that, the participants in the augmented group will receive 15-minutes of augmented music. After completion of the music, Study Staff will have the participants provide 1.5-2mL of saliva and remove the HR belt. Following removal of the HR belt, the participants will complete the post-survey.
  Interventions: Behavioral: Augmented Theme
- Mozart Theme (Active Comparator): In phase 2:
  Participants complete the pre-survey, and provide 1.5-2mL of saliva. Then, they will be equipped with a HR band (polar exercise band). After that, the participants will receive 15-minutes of the control music featuring a Mozart composition. After completion of the music, Study Staff will have the participants provide 1.5-2mL of saliva and remove the HR belt. Following removal of the HR belt, the participants will complete the post-survey.
  Interventions: Behavioral: Mozart Theme

INTERVENTIONS:
Behavioral: Augmented Theme — The music is augmented by embedding the natural rhythms of bodily functions (e.g. breathing, heart rate variability, vascular tone, etc) that signal the body to calm.
  Arms: Augmented Theme
Behavioral: Mozart Theme — The selected Mozart composition consists of: Composition Eine kleine Nachtmusik, K. 525 (5 minutes 30 seconds), Andante from Piano Concerto No. 21, K. 467 (6 minutes 30 seconds), and Ave verum corpus, K. 618 (3 minutes).
  Arms: Mozart Theme

SUMMARY:
The goal of this clinical trial is to explore possible benefits and mechanisms through which listening to music can improve health and wellness. The main goals of the study are:

* To investigate whether pre-survey measures of autonomic reactivity relate to the overall functioning of participants.
* To examine the immediate effects of listening to the augmented music.
* To identify individual characteristics that influence the immediate effects of listening to the augmented music.

Participants will:

PHASE 1:

* Complete the online pre- and post-surveys
* Listen to the brief music demo
* Listen to the full 15-minutes music session

PHASE 2:

* Complete the online pre- and post-surveys.
* Heart rate data will be collected continuously for about 25 minutes. It will be collected for 5 minutes before and after the intervention, and for 15 minutes during the intervention.
* Provide pre- and post- music saliva samples (1.5mL).
* Listen to full 15-minutes music session.

DETAILED DESCRIPTION:
The purpose of the current study is to explore the effects of listening to 15-minutes of sonic augmented music on subjective feelings of calmness and autonomic state.

Specific Aims:

Specific Aim 1: To investigate whether pre-intervention measures of ANS reactivity relate to the overall functioning of the participants.

•The investigators will examine measures of autonomic reactivity to prior mental health and medical adversity, embodiment, and emotional and physical health.

Specific Aim 2: To identify the immediate effects of listening to the music

•The investigators will explore whether listening to the music leads to improvements in the functioning. First, the investigators will compare the participants who opted to leave after the brief music demonstration to the participants who stayed for the additional 15-minutes of music. Next, the investigators will focus on improvements following listening to the music.

Specific Aim 3: To identify individual characteristics that influence the effectiveness of listening to the music immediately

•The investigators will explore the impact of specific vulnerability and resiliency factors (e.g., prior mental and medical adversity) on how well participants benefit from listening to the music immediately.

Specific Aim 4: To investigate levels of oxytocin and HRV after listening to calming music.

•The investigators will explore whether listening to music leads to changes in physiological and emotional responses, focusing on oxytocin as a marker of stress response. Specifically, we will compare the levels of salivary oxytocin before and after the intervention in two groups: participants who listen to 15 minutes of the Mozart theme and participants who listen to 15 minutes of the augmented theme. We will also measure heart rate (HR) using a wearable HR monitor to assess autonomic nervous system functioning and determine whether changes in HR are associated with changes in oxytocin levels following the music intervention. (Phase 2 only)

Experimental design

PHASE 1:

* Participation is limited to those attending the online workshop
* The participants will complete pre- and post-assessments that involve online measures.
* Music will be provided first in a brief music demo and then again in a 15-minute session.
* Between-subject analyses will compare those who listened only to the brief demo and withdrew participation against those who remained and listened to the 15-minutes of music to determine if those who listened to the 15-minutes of music exhibit greater improvements than those who did not. Within-subject analyses will determine the potential benefits of listening to the music for all participants.

PHASE 2:

* The participants will be randomly assigned to either the augmented music group or the control group featuring a Mozart composition.

  * Augmented music group: The music is augmented by embedding the natural rhythms of bodily functions (e.g. breathing, heart rate variability, vascular tone, etc) that signal the body to calm.
  * Control group: The selected Mozart composition consists of: Composition Eine kleine Nachtmusik, K. 525 (5 minutes 30 seconds), Andante from Piano Concerto No. 21, K. 467 (6 minutes 30 seconds), and Ave verum corpus, K. 618 (3 minutes). This composition is structured to serve as emotionally immersive, musically coherent control conditions in a 15-minute experimental paradigm.
* The control group will listen to 15 minutes of control music, and the augmented group will listen to 15 minutes of augmented music.
* At pre- and post-, the participants will complete online self-report surveys and provide 1.5mL of saliva.
* Heart rate data will be collected continuously for about 25 minutes. It will be collected for 5 minutes before and after the intervention, and for 15 minutes during the intervention. Markers will inserted to later separate the data into segments representing the 5 minutes before the music (baseline), time during the music, and 5 minutes after the administration of the music.
* Between-subject analyses will compare those who listened only to the augmented 15-minute music sample and those who listened to the control 15-minutes of music to determine if those who listened to the augmented music exhibit greater changes than those who did not. Subject analyses will determine the potential benefits of listening to music for all participants.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Between the ages of 18 and 89
* Proficient in English
* Attendees of an online workshop session

Exclusion Criteria:

- Over the age of 89

Phase 2:

Inclusion Criteria:

* Between the ages of 18 and 45
* Proficient in English

Exclusion Criteria:

- Over the age of 45

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Assessing the Impact of Autonomic Reactivity using the Body Perceptions Inventory Short Form | Baseline
  This 20-item measure is scored on a 5-point Likert scale (never = 1, occasionally = 2, sometimes = 3, usually = 4, always = 5). Items are summed to determine total autonomic reactivity score, with the higher scores indicating greater autonomic reactivity
Assessing the Impact of Adversity History on the Effectiveness of Listening to Music | Baseline
  This measure assesses the impact of six types of traumatic experiences (childhood adverse experiences, childhood maltreatment, intimate partner maltreatment, other person maltreatment, life-threatening situations, sudden losses, and person health situations). Each item is scored on a 5-point Likert scale (did not occur = 0, occurred and no impact on my life = 1 to big impact on my life = 4). Items are summed to determine total impact scores.
Measuring Change in subjective feelings of calmness and autonomic state using the Benefits List | From baseline through study completion, an average of 90 minutes
  This 20-item measure, which assesses subjective feelings of calmness and autonomic state was created for this study.
Assessing the Impact of anxiety on the Effectiveness of Listening to Music using the GAD-7 | Baseline
  This 7-item measure assesses the severity of generalized anxiety symptoms. It is scored on a 4-point Likert scale (not at all = 0, several days = 1, more than half the days = 2, nearly every day = 3). The items are summed to calculate the total anxiety score, with higher scores indicating more severe anxiety symptoms.
Assessing the Impact of depression on the Effectiveness of Listening to Music using the PHQ-8 | Baseline
  This 8-item measure assesses the severity of depressive symptoms. It is scored on a 4-point Likert scale (not at all = 0, several days = 1, more than half the days = 2, nearly every day = 3). The items are summed to determine the total depression score, with higher scores indicating greater severity of depressive symptoms.
Assessing the Impact of loneliness on the Effectiveness of Listening to Music using the UCLA Loneliness | Baseline
  This 20-item measure assesses how often a person feels disconnected from others. It is scored on a 4-point Likert scale (never = 1, rarely = 2, sometimes = 3, often = 4). The items are summed to calculate the total loneliness score, with higher scores indicating greater feelings of loneliness.
Assessing the Impact of hostility on the Effectiveness of Listening to Music using the Cook-Medley | Baseline
  This 60-item measure assesses the level of hostility and negative affectivity. It is scored on a true/false format, where responses are recorded as 1 for "true" and 0 for "false." The items are summed to determine the total hostility score, with higher scores indicating greater levels of hostility.
Assessing the Impact of cardiovascular risk on the Effectiveness of Listening to Music using the QRISK3 | Baseline
  The QRISK3 is a risk assessment tool used to estimate the 10-year risk of developing cardiovascular disease. It is based on a variety of factors, including age, sex, blood pressure, cholesterol levels, smoking status, and medical history. The score is calculated using a point-based system, with higher scores indicating a higher risk of cardiovascular events. The result provides an estimated percentage of risk over the next 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes P Dale, PhD, Principal Investigator — University of Florida; John P Williamson, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida McKnight Brain Institution, Gainesville, Florida
  - UF Health Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to protect the privacy of participants.